CLINICAL TRIAL: NCT06029738
Title: The Effect on Obsessive-Compulsive Beliefs and Symptoms of Metacognition Training Given to Patients With Obsessive Compulsive Disorder (MCT-OCD)
Brief Title: Effect on Obsessive-Compulsive Beliefs and Symptoms of MCT-OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zeynep Koc, Research Assistant, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethics Protocol Code: 2022/13
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive Symptoms; Compulsive Symptoms; Obsessive Beliefs; Compulsive Beliefs; Obsessive-Compulsive Disorder; OCD; Metacognitive Training for Obsessive-Compulsive Disorder; MCT-OCD; Randomized Controlled Trial; RCT
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The research was planned as two groups randomized controlled trial study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Intervention (Metacognitive Education for Obsessive-Compulsive Disorder (MCT-OCD)): MCT-OCD is a group education for OCD patients
  Interventions: Behavioral: Metacognitive Training for Obsessive-Compulsive Disorder (MCT-OCD)
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Metacognitive Training for Obsessive-Compulsive Disorder (MCT-OCD) — MCT-OCD is a group education for OCD patients.
  Arms: Experimental group

SUMMARY:
Objective: Since Metacognitive Training for Obsessive-Compulsive Disorder (MCT-OCD) targets and interferes with dysfunctional (meta-)cognitive beliefs, metacognitions, cognitive biases and coping strategies that contribute to the development and maintenance of OC symptoms, it is predicted that MCT-OCD can be highly effective on obsessive-compulsive beliefs and symptoms. Therefore, this study aims to examine the effect of metacognitive training (MCT-OCD) given to patients with obsessive-compulsive disorder on obsessive-compulsive beliefs and symptoms.Type of Study: The study was planned as a single-blind randomized controlled trial study. Dependent and Independent Variables of the Research: Dependent Variables: Padua Inventory, Obsessive Beliefs Scale and Beliefs About Rituals Scale mean scores. Independent Variables: Metacognitive Training for Obsessive-Compulsive Disorder. Control Variables: Age, gender, marital status, educational status, medicine use, and hospitalization history. Place of Research: The research will be conducted in the Psychiatry Polyclinic of Gaziantep University Şahinbey Research and Application Hospital in Gaziantep City Center. Population and Sample of the Research: The population of the research will be the patients who received treatment with a diagnosis of OCD according to DSM-5 in the Psychiatry Outpatient Clinic of Gaziantep University Şahinbey Research and Application Hospital at the time of the study, and the sample will consist of individuals who meet the inclusion criteria of the study. In this study, a priori power analysis was performed by using the G Power 3.9.1 program to calculate the sample size. The studies were examined (Miegel et al. 2022) and the expected confidence intervals of the Obsessive Beliefs Scale were determined, while the confidence interval was α=0.05, the power of the test (1-β) was 0.80, the effect size was d=0.6630086, while the experimental group was 37 and the control group was 37. A total of 74 patients were calculated. Considering that there will be losses in the research, it is planned to study with 80 people (40 experimental and 40 control groups).

DETAILED DESCRIPTION:
Research Goals:

Goal-1: To determine the obsessive-compulsive beliefs of patients with obsessive compulsive disorder in the experimental and control groups Goal-2: To determine the obsessive compulsive symptom levels of patients with obsessive compulsive disorder in the experimental and control groups Goal-3: Reducing obsessive-compulsive beliefs of patients with obsessive compulsive disorder in the experimental group with the application of metacognitive training Goal-4: Reducing the symptom levels of patients with obsessive compulsive disorder in the experimental group with the application of metacognitive training Goal-5: It is aimed to create high-level evidence to reduce obsessive-compulsive beliefs and symptom level of patients with obsessive compulsive disorder.

Research Hypotheses:

H0: Metacognitive training given to patients with obsessive compulsive disorder has no effect on obsessive-compulsive beliefs and symptom levels of patients in the experimental and control groups.

H1a Hypothesis: Metacognitive training given to patients with obsessive compulsive disorder will decrease the mean obsessive belief scores of the patients in the experimental group compared to the patients in the control group.

H1b Hypothesis: Metacognitive training training given to patients with obsessive compulsive disorder will decrease the mean compulsive belief scores of the patients in the experimental group compared to the patients in the control group.

H1c Hypothesis: Metacognitive training given to patients with obsessive compulsive disorder will decrease the mean obsessive-compulsive symptom scores of the patients in the experimental group compared to the patients in the control group.

H2a: With the metacognitive training given to patients with obsessive compulsive disorder, obsessive beliefs mean scores of the patients in the experimental group will decrease after the intervention compared to the pre-intervention.

H2b: With the metacognitive training given to patients with obsessive-compulsive disorder, the mean scores of compulsive beliefs of the patients in the experimental group will decrease after the intervention compared to the pre-intervention.

H2c: With the metacognitive training given to patients with obsessive compulsive disorder, obsessive-compulsive mean scores of the patients in the experimental group will decrease after the intervention compared to the pre-intervention.

Type of Study: The study was planned as a single-blind Randomized controlled trial study.

Dependent and Independent Variables of the Research:

Dependent Variables: Padua Inventory, Obsessive Beliefs Scale and Beliefs About Rituals Scale mean scores.

Independent Variables: Metacognitive Training for Obsessive-Compulsive Disorder.

Control Variables: Age, gender, marital status, educational status, medicine use, and hospitalization history.

Place of Research: The research will be conducted in the Psychiatry Polyclinic of Gaziantep University Şahinbey Research and Application Hospital in Gaziantep City Center.

Population and Sample of the Research: The population of the research will be the patients who received treatment with a diagnosis of OCD according to DSM-5 in the Psychiatry Outpatient Clinic of Gaziantep University Şahinbey Research and Application Hospital at the time of the study, and the sample will consist of individuals who meet the inclusion criteria of the study. In this study, a priori power analysis was performed by using the G Power 3.9.1 program to calculate the sample size. The studies were examined (Miegel et al. 2022) and the expected confidence intervals of the Obsessive Beliefs Scale were determined, while the confidence interval was α=0.05, the power of the test (1-β) was 0.80, the effect size was d=0.6630086, while the experimental group was 37 and the control group was 37. A total of 74 patients were calculated. Considering that there will be losses in the research, it is planned to study with 80 people (40 experimental and 40 control groups). Participants included in the study will be assigned to the experimental and control groups by simple randomization in the computer environment. If the number of people who leave the study for various reasons is high, the intervention may seem less effective than it is. All individuals included in randomization should be included in the analysis in order to evaluate the effectiveness of the intervention. Whittaker et al. (2006). For this reason, intention to treat (ITT) analysis will be performed as a lost data analysis when sample loss (in case of more than 20% predicted) is experienced in randomized controlled studies. The ITT analysis enables individuals in the intervention and comparison groups to be compared in the groups to which they were randomly assigned.

Randomization: Randomization was performed using the randomization list Medcalc version 18.11.3, for the assignment of patients to groups. Patients who were referred by the polyclinic doctor, met the inclusion criteria, and agreed to participate in the study will be numbered in the order of their referral. The correspondence of the number received by the patient at the end of the randomization list obtained from Medcale will determine whether the patient is in the experimental or control group. Patients will not know which group they are in. Thus, the research will be done with a single blind. Randomization and working process will be shown in the 2010 CONSORT Flowchart (http://www.consort-statement.org/consort-statement/flow-diagram).

Data Collection Tools: As a data collection tool in this research; Personal information form prepared by the researcher, Padua Inventory-Washington State University Revision (PE-WEÜR) to evaluate OCD symptoms, Obsessive Beliefs Scale (OBS) to measure beliefs about obsessions, and Beliefs About Rituals Scale (BIAS) for beliefs about Compulsions will be used.

Application of Research The research will be carried out in two stages, namely preparation and implementation. Preparation phase: Collaboration with the team in the polyclinic where the research will be conducted will be provided and Metacognitive Training for Obsessive-Compulsive Disorder (MCT-OCD) will be published as a booklet. Implementation phase: determining the target sample group, randomly forming the experimental and control groups, and applying the Metacognitive Training for Obsessive-Compulsive Disorder to the experimental group will include the evaluation stages of the application results.

Preparation Phase of the Research:

Establishing suitable conditions for the research by cooperating with the team in the polyclinic where the research will be conducted: Meeting with the team in the polyclinic where the research will be conducted, information will be provided and cooperation will be provided, and the room where the training will be held will be arranged.

Publishing of Manual of The Metacognitive Training for Obsessive-Compulsive Disorder: In order to increase the competence of the researcher who will make the application, he successfully completed and was entitled to receive a certificate the 50-hour cognitive and behavioral therapy theoretical training and the 30-hour CBT skill acquisition and supervision practice training given by the Cognitive Behavioral Psychotherapies Association. Since the Metacognitive Training for Obsessive-Compulsive Disorder has no translation into Turkish, it is planned to translate this research during the preparation process. For this purpose, permission was obtained from the developers of the training/Clinical Neuropsychology Working Group via e-mail and the content of the training was provided in order to use the MCT-OCD initiative and to make its Turkish translation and version. After the Turkish translation and version of each module of the training were made, it was sent to the developers. The requested corrections were made until the Turkish version and translation of each submitted module was approved. Thus, approval was obtained for the final version of the presentation and homework of each module. In this process, after all the modules of MCT-OCD were translated, the Turkish translation and version were brought to the literature by us as MKE-OKB and published on the Clinical Neuropsychology homepage and made available for free. The educational content published in this process will be published as a booklet. This booklet will be distributed to the patients in the experimental group at the beginning of the training, and to the patients in the control group after the follow-up test.

Application Phase of the Research: During the implementation phase of the study, patients with a diagnosis of OCD will be directed to the researcher by the polyclinic doctor. Referred patients will be evaluated in terms of inclusion criteria. Patients who meet the inclusion criteria will be informed about the study. After the information, the patients who accepted to participate in the study will be randomized according to the randomization list and group assignment will be made. If the randomized patient is assigned to the control group, the patient will be informed about the research process, the frequency of the survey, and an informed consent form prepared for the control group will be signed. If the patient is assigned to the experimental group, the patient will be informed about the research process, MCT-OCD and the education process, and an informed consent form prepared for the experimental group will be signed. The training days and hours of the patient will be determined. A face-to-face evaluation interview will be conducted for the patients in the experimental and control groups just before the training to administer the pre-tests (Personal Information Form, Padua Inventory-Washington State University Revision (PE-WEUR), Obsessive Beliefs Scale (OBS), Beliefs About Rituals Scale (BRS). Training will be conducted in a group format with face-to-face interview technique. Each group and session will include 3-10 OCD patients. MCT-OCD group sessions will be conducted by the researcher, who has received CBT therapy training and is a psychiatric nursing doctoral student. Metacognitive training consisting of 8 modules will be given to the patients in the experimental group, It will be applied once a week in the form of 1 module. Each session of the metacognitive training will last for a total of 90 minutes, 45+45 (break in between). Before the training, the patients will be called by phone and the training time will be reminded. To make it easier for the patients to apply the knowledge and skills they have acquired from MCT-OCD to their daily lives Each patient will be given a booklet with a summary of all modules, homework and exercises at their first session.

Intervention (Metacognitive Education for Obsessive-Compulsive Disorder (MCT-OCD)): MCT-OCD is a group education for OCD patients (Jelinek et al. 2018). MCI-OCD is in an open group format that allows patients to join the group at any time (all patients complete all modules but can start with a different module) (Miegel et al. 2020a, 2021). MCT-OCD consists of highly standardized slide-based multimedia presentations (Miegel et al. 2021). MCT-OCD is based on a self-help manual, myMCT (Moritz & Hauschildt, 2016). TCI-OCD includes some elements from cognitive behavioral therapy, but mainly focuses on cognitive biases and metacognitions related to OCD. The revised version of MCT-OCD consists of eight modules aiming to change patients' dysfunctional (meta-) cognitive beliefs, prejudices and dysfunctional coping strategies: (1) myths about OCD; (2) perfectionism (with additional slides on stigma); (3) intolerance to uncertainty (with additional slides on depression); (4) fusion beliefs (with additional slides on self-worth); (5) control of thoughts; (6) exaggeration of the threat (with additional slides on rumination); (7) exaggerated responsibility and (8) biased attention and cognitive networks. (Miegel et al., 2020a, 2023b). In all modules, the related dysfunctional process concept is first introduced, then newer and functional coping strategies are proposed to deal with various dysfunctional (meta-) cognitive beliefs, prejudices and dysfunctional coping strategies (Miegel et al. 2020a). The contents of each module are listed as follows: The term "metacognition" and the purpose of TCI-OCD are explained only if it is the patient's first MCT-OCD session; homework is discussed; the targeted (meta-) cognitive belief is introduced in the session; Examples and exercises related to (meta-)cognitive belief are provided; functional coping strategies are introduced; the content covered in the module is summarized; closure is done with the opportunity to share what the patients have learned (Miegel et al. 2023b). Detailed content of all modules of MKE-OCD is available in Table-1. In addition, the content of all modules of MKE-OKB, the Turkish version of MCT-OCD, can be accessed at https://clinical-neuropsychology.de/mct-ocd-turkish/.

Application of post-tests and follow-up tests to the experimental and control groups: Immediately after the completion of the Metacognitive Training sessions, the post-test will be applied to the patients in the experimental group and the follow-up test will be applied 3 months after the post-test application. In the control group, no intervention will be made and the follow-up test will be applied 8 weeks after the pre-test and 3 months after the post-test. After the follow-up test is applied, the control group will be given a training booklet prepared in line with the content of the program.

Evaluation of Data: Statistical analyzes of the research will be made using the SPSS 22 package program. The normal distribution of the data will be evaluated by Kolmogrov Smirnov tests, Skewness and Kurtosis values. Parametric tests will be used to evaluate the data that fit the normal distribution. In the evaluation of the data, percentage, arithmetic mean and standard deviation will be used in the distribution of the descriptive characteristics of the patients in the experimental and control groups. In cases where the assumption of normal distribution is provided in the analysis of the data, the independent sample t-test is used to compare the means of two independent groups in the comparison of quantitative data; In cases where the normal distribution assumption is not met, the Mann Whitney U test will be used. In the comparison of the mean of more than two independent groups, ANOVA will be used for tests with normal distribution, and Kruskal Wallis H test will be used for data that are not normally distributed. In order to determine the difference in the results with difference, multiple comparison test will be done. Chi-square analysis will be done to examine the relationship in categorical data. For the analysis of repeated measurements, in cases where the assumption of normal distribution is provided, ANOVA for repeated measurements; In cases where the assumption of normal distribution is not satisfied, the Friedman test will be used. In all analyzes, the confidence interval will be 95% and the significance will be considered as p<0.05.

Ethical Principles of the Study: Approval was obtained from the Gaziantep University Clinical Research Ethics Committee in order to conduct the study (Protocol code: 2022/13). Written and verbal permission was obtained from the center where the research would be conducted. The research will be conducted in accordance with the Declaration of Helsinki. During the collection of research data, individuals will have to sign an "Informed Consent Form" about the research. The principle of "Respect for Autonomy" will be followed by stating that they are free to participate in the research and to leave whenever they want after participating in the research, and the principle of "Confidentiality and Protection of Confidentiality" will be fulfilled by stating that the information of the patients participating in the research will be kept confidential.

Reporting the Research: CONSORT 2010 guidelines will be followed in the conduct and reporting of the research, checklist and flowchart will be used (Schulz et al. 2010; Moher et al. 2012; http://www.consort-statement.org)

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study, Not having a condition that prevents communication, Being between the ages of 18-65, Being followed up with the diagnosis of OCD (Obsession-Compulsive Disorder) according to DSM-5 criteria; Being literate; Not being included in such a training program for the disease in the last 5 years.

Exclusion Criteria:

* Those diagnosed with another comorbid mental illness; Patients with mental disorders such as intellectual disability or dementia that makes it impossible to cooperate; Patients who are illiterate; Patients who do not consent for the interview.

Expulsion Criteria:

* Patients in the experimental group who want to quit the study during the study period and who do not attend at least two modules/sessions of the training are within the scope of the exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Padua Inventory mean scores | 0-2-5. months
  PEWEUR is a 39-item self-report scale that evaluates obsessions and compulsions. The Padua Inventory was developed by Sanavio (1988) and Burns et al. (1996) made the PE-WEÜR version. The Turkish validity study of the scale was conducted by Yorulmaz et al. (2007) made by and. The scale is in a five-point Likert type, ranging from 0 = Not at all to 4 = Very much. In scoring the scale, each sub-dimension is scored within itself. The high score obtained from each sub-dimension of the scale indicates that the individual's anxiety level evaluated by the relevant sub-dimension is high. In the Turkish validity and reliability study, PI-WEÜR consists of 5 sub-dimensions: Obsessions and compulsions of checking; Dirty obsessions and cleaning compulsions, Obsessive urges to harm others/self; Regulation, Obsessive thoughts of harming others/self. The cronbach α value of the scale was found to be 0.93 (Yorulmaz et al. 2007).
Obsessive Beliefs Scale mean score | 0-2-5. months
  Obsessive Beliefs Scale (AS-44): OBS-44 was developed to identify key cognitions in OCD, consisting of three subscales (exaggerated sense of responsibility/danger expectation, perfectionism/need for certainty, giving importance to thoughts/controlling thoughts). The need for self-report) is a 44-item self-report scale with each item scored between 1 and 7, with higher scores indicating greater belief in those cognitions (OCCWG, 2005). Cut-off scores for this scale were not reported. The Turkish version of the SPQ was also found to be valid and reliable. Boysan et al. (2010) conducted a Turkish validity study and the cronbach α was found to be 0.95.
Beliefs About Rituals Scale mean scores | 0-2-5. months
  Beliefs About Rituals Scale (BRS): BRS is a 12-item self-report scale that evaluates beliefs about rituals and consists of three subscales (behavior and character change, guilt and loss of functionality, anxiety). Scale items are scored between 1-4. In the scale, a description of the rituals is given first, followed by an example, and the participants are asked what they believe will happen if this ritual is not performed. High scores indicate a high number of beliefs (undesirable character and behavior changes, guilt and loss of functionality, anxiety) that performing rituals prevents the feared consequences. There is no cutoff score. In the original validity and reliability study of the scale, the Cronbach α value was found to be 0.82 (McNicol & Wells, 2012). The Turkish validity study of the scale was conducted by Güneysu et al. (2020) and Cronbach α = 0.856 was found.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Koç, MsC, Principal Investigator — University of Gaziantep; Derya Tanrıverdi, Prof.Dr., Study Director — University of Gaziantep

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miegel F, Cludius B, Hottenrott B, Demiralay C, Sure A, Jelinek L. Session-specific effects of the Metacognitive Training for Obsessive-Compulsive Disorder (MCT-OCD). Psychother Res. 2020 Apr;30(4):474-486. doi: 10.1080/10503307.2019.1613582. Epub 2019 May 9. PMID 31072282
- [Background] Miegel F, Demiralay C, Moritz S, Wirtz J, Hottenrott B, Jelinek L. Metacognitive Training for Obsessive-Compulsive Disorder: a study protocol for a randomized controlled trial. BMC Psychiatry. 2020 Jul 6;20(1):350. doi: 10.1186/s12888-020-02648-3. PMID 32631261
- [Background] Miegel F, Rubel J, Ching THW, Yassari AH, Bohnsack F, Duwe M, Jelinek L. How to assess and analyse session-specific effects and predictors: An example with the Metacognitive Training for Obsessive-Compulsive Disorder intervention. Clin Psychol Psychother. 2023 Sep-Oct;30(5):1158-1169. doi: 10.1002/cpp.2876. Epub 2023 Jun 8. PMID 37288873
- [Background] Obsessive Compulsive Cognitions Working Group. Psychometric validation of the obsessive belief questionnaire and interpretation of intrusions inventory--Part 2: Factor analyses and testing of a brief version. Behav Res Ther. 2005 Nov;43(11):1527-42. doi: 10.1016/j.brat.2004.07.010. PMID 16299894
- [Background] Burns GL, Keortge SG, Formea GM, Sternberger LG. Revision of the Padua Inventory of obsessive compulsive disorder symptoms: distinctions between worry, obsessions, and compulsions. Behav Res Ther. 1996 Feb;34(2):163-73. doi: 10.1016/0005-7967(95)00035-6. PMID 8741724
- [Background] Sanavio E. Obsessions and compulsions: the Padua Inventory. Behav Res Ther. 1988;26(2):169-77. doi: 10.1016/0005-7967(88)90116-7. No abstract available. PMID 3365207
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- See also: CONSORT 2010, Erişim Tarihi: 28.08.2023. — http://www.consort-statement.org